CLINICAL TRIAL: NCT06296095
Title: A Single-center, Single-arm, Open-label, Dose-escalation Clinical Study Evaluating the Safety, Tolerability, and Initial Efficacy of CUD005 Injection in Patients With Cirrhosis
Brief Title: To Evaluate the Clinical Study of CUD005 Injection in Patients With Cirrhosis
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KDS-CUD-1
Record Dates: First submitted 2023-07-17; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Cirrhosis, Liver
Keywords: Cirrhosis; cell therapy; PBMC; safety; tolerability; MTD; DLT; dose escalation
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): cell therapy
  Interventions: Biological: Cell therapy

INTERVENTIONS:
Biological: Cell therapy — Subjects were placed sequentially into three different dose groups, 5.0×107 cells/time (low-dose group), 1.5×108 cells/time (medium-dose group), and 5.0×108 cells/time (high-dose group) for dose escalation

SUMMARY:
The study is a single-center, single-arm, open-label, dose-escalation clinical study, to evaluate the tolerability, safety and preliminary efficacy of CUD005 injection in patients with cirrhosis

DETAILED DESCRIPTION:
The study was designed according to the 3+3 principle, with a total of 3 dose levels and dose escalation.

Low-dose group: 5.0×107 cells/time; Medium-dose group: 1.5×108 cells/time; High-dose group: 5.0×108 cells/time. Subjects were sequentially placed in 3 different dose groups administered as a single peripheral intravenous dose.

According to the enrollment restriction design, a total of a minimum of 9 subjects are expected to be enrolled, and the final sample size depends on the number of DLT, the number of dose groups ascended before DLT is observed, and the MTD is determined.

ELIGIBILITY:
Inclusion Criteria:

1. BMI≤30 kg/m2
2. The results of liver histopathological examination were consistent with the Ishak stage of liver fibrosis ≥3 points；
3. Consent to liver histopathological examination before and after cell therapy (The subject is exempted from liver histopathological examination during the screening period, if he has been performed liver histopathological examination within 2 months before signing the informed consent)；
4. Subjects were able to communicate well with the investigator, cooperate with follow-up work, and understand and comply with the requirements of the study.

Exclusion Criteria:

1. Subjects who were Allergic to cell therapy, steroids, and related drugs used in the study；
2. Have malignant tumors, history of organ transplantation or tissue regeneration therapy, active, known or suspected autoimmune diseases, idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, active pneumonia, heart disease that is not well controlled, hypertension, etc;
3. Subjects with stage III or IV hepatic encephalopathy within 3 months before apheresis or currently diagnosed；
4. Virology shows anti-HCV antibodies, HIV-positive, or syphilis antibodies during the screening period；
5. Subjects were HBV surface antigen positive and HBV-DNA titer was ≥ 20 IU/mL during the screening period；
6. Subjects with clinically symptomatic ascites or pleural effusions requiring puncture drainage. Or who had received thoracic and ascites drainage within 2 weeks prior to treatment, had may only show a small amount of ascites or pleural effusions on imaging, except in those without clinical symptoms；
7. According to the judgment of the investigator, the subjects had other factors that may cause the study to be terminated halfway, such as other serious concomitant diseases (such as severe diabetes, mental illness, drug use, etc.), serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT,MTD | 28 days
  Dose-limiting toxicity（DLT）: frequency of occurrence, level of dose of DLT toxicity;Maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
fibrosis staging and inflammatory grading | 180 days
  Histological changes in liver biopsy at day 180 after cell therapy.Methods: A small amount of liver tissue was taken from the liver by percutaneous puncture, and its histological changes were observed directly under the microscope. According to the pathological results, the Ishak scoring system for liver fibrosis (which includes fibrosis stage and inflammation grade evaluation criteria) was used to evaluate liver fibrosis, in which 0 was the best and 6 was the worst.
All-cause mortality | 1 year
  the ratio of the total number of deaths due to various factors over 1 year of cell therapy to the number of people in this population for the same period
TE（Transient elastography） | 1 year
  Changes in transient elastography.Methods: A special probe was used to generate an instantaneous low-frequency pulse to cause instantaneous displacement and shear wave in the liver tissue. The shear wave was tracked and collected to obtain the elastic modulus of the tissue, and the degree of liver fibrosis was evaluated by liver stiffness measurement (LSM). The higher the shear wave velocity, the higher the LSM value, and the stiffer the liver tissue in the detection area.

OTHER OUTCOMES:
MELD（Model for End-stage Liver Disease） | 1 year
  Changes in the Model of End-Stage Liver Disease.Methods: Creatinine, international normalized ratio (INR), and bilirubin combined with the etiology of liver cirrhosis were used to evaluate liver function reserve and prognosis in patients with chronic liver disease. Formula: MELD=3.78×ln [T-BiL(mg/dl)]+11.2×ln[INR]+9.57×ln[Cr (mg/dl)]+ 6.43× cause (0 for cholestatic and alcoholic cirrhosis, 1 for cirrhosis due to other causes such as viruses)

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin LX Liu, Professor, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui province hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No